CLINICAL TRIAL: NCT02250378
Title: Feasibility Study of Stereotactic Body Radiation Therapy Followed by Wedge Resection for Peripherally Located Early Stage Non-small Cell Lung Cancer
Brief Title: Stereotactic Radiosurgery Followed by Wedge Resection in Treating Patients With Early Stage Peripheral Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2N-14-3; NCI-2014-01916 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2N-14-3 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IA Non-small Cell Lung Cancer; Stage IB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (stereotactic radiosurgery, wedge resection) (Experimental): Patients undergo stereotactic radiosurgery every other day for 3 or 5 fractions (depending on the size tumor and proximity to the chest wall). Within 4-6 weeks after completion of stereotactic radiosurgery, patients undergo wedge resection.
  Interventions: Radiation: stereotactic radiosurgery; Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Other: quality-of-life assessment

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Undergo stereotactic radiosurgery
Procedure: therapeutic conventional surgery — Undergo wedge resection
Other: laboratory biomarker analysis — Correlative studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies the side effects and how well stereotactic radiosurgery followed by wedge resection works in treating patients with early stage non-small cell lung cancer that is located in the outer, or peripheral, areas of the lung. Stereotactic radiosurgery, also known as stereotactic body radiation therapy, is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Wedge resection is a less invasive type of surgery for removal of the tumor and a small amount of normal tissue around it. Giving stereotactic radiosurgery followed by wedge resection may be a safe treatment option for patients who cannot receive standard treatment with lobectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of a wedge resection following stereotactic body radiation therapy (SBRT) for early stage peripheral non-small cell lung cancer (NSCLC).

SECONDARY OBJECTIVES:

I. To assess pathologic response rates to SBRT as determined by pathologic examination of resected tumors.

II. To prospectively assess patient quality of life when treated with SBRT and wedge resection.

TERTIARY OBJECTIVES:

I. To describe the location of viable tumor and to correlate pathologic response rates with radiation dose, size of tumor, and tumor histology.

II. To correlate pathologic response rates and functional imaging with pre- and post-treatment dual-input perfusion (DP)-computed tomography (CT) and positron emission tomography (PET)-CT.

III. To correlate changes in serum levels of deoxyribonucleic acid (DNA) methylation and circulating tumor cells (CTC) with pathologic response rates.

OUTLINE:

Patients undergo stereotactic radiosurgery every other day for 3 or 5 fractions (depending on the size tumor and proximity to the chest wall). Within 4-6 weeks after completion of stereotactic radiosurgery, patients undergo wedge resection.

After completion of study treatment, patients are followed up at 1, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Biopsy proven non-small cell lung cancer
* Maximum tumor dimension =< 5 cm
* No clinical evidence of N1, N2 or N3 lymph nodes as assessed by CT and/or PET-CT
* No evidence of distant metastatic disease
* Tumor verified by a thoracic surgeon to be in a location that will permit a sublobar resection
* Tumor located peripherally within the lung (peripheral defined as not touching any surface within 2 cm of the proximal bronchial tree in all directions) and not touching the mediastinal pleura
* Pulmonary function tests (PFTs) with diffusing capacity of the lung for carbon monoxide (DLCO) within 90 days prior to registration
* Patient at high-risk of complications from lobectomy meeting a minimum of one major criteria or two minor criteria as described below:

  * Major criteria

    * Predicted postoperative forced expiratory volume in one second (FEV1) =< 40%
    * Predicted postoperative DLCO =< 40%
    * Age >= 72
  * Minor criteria

    * Predicted postoperative FEV1 41-60%
    * Predicted postoperative DLCO 41-60%
    * Pulmonary hypertension (defined by a pulmonary artery systolic pressure greater than 40 mm Hg) as estimated by echocardiography or right heart catheterization
    * Poor left ventricular function (defined as an ejection fraction 40% or less)
    * Resting or exercising arterial partial pressure of oxygen (pO2) =< 55 mmHg or oxygen saturation (SpO2) =< 88%
    * Partial pressure of carbon monoxide (pCO2) > 45 mm Hg
    * Modified Medical Research Council Dyspnea Scale >= 3
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

  * A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Pregnant women
* Patients with central tumors within the proximal tree or touching the mediastinal pleura
* Patients with evidence of distant metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Rate of grade 3-5 adverse events, graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 12 months after surgery
  Treatment related toxicities will be assessed and recorded for each patient receiving treatment.
Rates of perioperative complications including blood loss, days in the intensive care unit, and operative time | Up to 12 months after surgery
Feasibility, determined by the number of patients who are able to complete wedge resection as well as receive the full dose of stereotactic radiosurgery | Up to 12 months after surgery

SECONDARY OUTCOMES:
Pathologic response rates | Up to 12 months after surgery
  The pathologic response rates will be determined by measuring the percent of viable cells in the resected specimen. Associations (e.g. between pathologic response rates and DP-CT, fludeoxyglucose [FDG] uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).
Quality of life assessment | Up to 12 months after surgery
  Quality of life assessments will be summarized over time with descriptive statistics.

OTHER OUTCOMES:
Imaging characteristics that may predict response based on DP-CT and PET-CT scans | Up to 30 days after stereotactic radiosurgery
  Associations (e.g. between pathologic response rates and DP-CT, FDG uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).
Changes in perfusion using DP-CT scans | Baseline to up to 30 days after stereotactic radiosurgery
  Changes in DP-CT will be compared between pre- and post-stereotactic radiosurgery scans to determine if changes in perfusion correlates with pathologic response. Associations (e.g. between pathologic response rates and DP-CT, FDG uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).
Changes in FDG uptake | Baseline to up to 12 months after surgery
  Changes in FDG uptake will be compared between pre- and post-SBRT scans to determine if changes in FDG uptake correlates with pathologic response. Associations (e.g. between pathologic response rates and DP-CT, FDG uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).
Changes in DNA methylation analysis | Baseline to up to 12 months after surgery
  The amount of DNA methylation in the blood as well as relative changes in counts will be correlated with pathologic outcomes. DNA methylation will be summarized over time with descriptive statistics. Associations (e.g. between pathologic response rates and DP-CT, FDG uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).
Changes in CTC levels | Baseline to up to 12 months after surgery
  The amount of CTC in the blood as well as relative changes in counts will be correlated with pathologic outcomes. CTC levels will be summarized over time with descriptive statistics. Associations (e.g. between pathologic response rates and DP-CT, FDG uptake, DNA methylation, and CTC levels) will be displayed visually with scatterplots or contingency tables and appropriate measure of association (Wilcoxon test, Fisher's exact test, Spearman correlation coefficient, and McNemar's test).

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Chung, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States